CLINICAL TRIAL: NCT01508429
Title: Misoprostol for the Treatment of Postpartum Haemorrhage (PPH) Following Self- Administration of Misoprostol Prophylaxis in Home Deliveries.
Brief Title: Misoprostol for Treatment of Postpartum Haemorrhage (PPH) in Home Births
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Aga Khan Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2.4.14
Record Dates: First submitted 2011-12-01; First posted 2012-01-12 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Postpartum Hemorrhage (PPH)
Keywords: Postpartum hemorrhage; PPH; misoprostol; home deliveries
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- misoprostol (Active Comparator): 800mcg misoprostol (four tablets of 200 mcg administered sublingually)
  Interventions: Drug: Misoprostol
- placebo (Placebo Comparator): 4 placebo tablets (resembling misoprostol) administered sublingually
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — 4 placebo tablets (resembling misoprostol) administered sublingually
  Arms: placebo
Drug: Misoprostol — 800mcg misoprostol (4 200mcg tablets administered sublingually)
  Arms: misoprostol

SUMMARY:
Misoprostol, a prostaglandin E1 that induces uterine contractions, has been proposed as a low cost, easy-to-use option for prevention and treatment of Postpartum Haemorrhage (PPH), especially in settings where injectable uterotonics are not yet available or feasible to use.

A double-blinded individual randomized controlled study of misoprostol versus placebo in home deliveries in four districts in the Badakshan Province in Afghanistan. The study will recruit pregnant women who are likely to deliver at home. All women enrolled in the study will receive 600 mcg misoprostol to be self-administered as prophylaxis for PPH after delivery of their baby (ies) and before delivery of the placenta.

Women who experience a PPH will be randomized to receive either: a) standard of care + 800 mcg misoprostol (four 200 mcg tablets) or b) standard of care + four placebo tablets resembling misoprostol. In this setting, standard of care is referral.

ELIGIBILITY:
Inclusion Criteria:

* Women must be pregnant
* Must be able to provide informed consent
* Must agree to have a community health worker present at the time of delivery
* Must agree to participate in a follow up interview by the study midwife
* Must agree to have pre and postpartum haemoglobin taken

Exclusion Criteria:

* Women who do not meet the inclusion criteria

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Hb of greater than or equal to 2 g/dl from pre- to post-delivery | 3-5 days after delivery
  The primary outcome will measure the proportion of women who experience a drop in their haemoglobin concentration (Hb) of greater than 2 g/dl from pre- to post-delivery. The outcome will be compared between the two treatment groups.

SECONDARY OUTCOMES:
Side effects | immediately after delivery; 3-5 days post delivery
  Observed side effects: perceived severity, additional care provided Any serious adverse outcomes including uterine rupture, hysterectomy, hospitalization, maternal deaths, and neonatal deaths.
additional interventions | immediately after delivery; 3-5 days post delivery
  Additional interventions and additional care provided to the woman, # of referrals and transfers
Acceptability | immediately after delivery; 3-5 days post delivery
  Acceptability and management of side effects, acceptablity of taking the drugs

CONTACTS AND LOCATIONS:
Overall Officials: Shafiq Mirzazada, Principal Investigator — Aga Khan Health Services; Gijs Walraven, Study Director — Secretariat of His Highness the Aga Khan, Aiglemont; Dina Abbas, Study Director — Gynuity Health Projects; Jill Durocher, Study Director — Gynuity Health Projects
Locations (1):
- Home delivery setting, Darwaz, Ishkashim, Shugnan, Wakhan Districts, Badakshan Province, Afghanistan

REFERENCES:
- [Derived] Parry Smith WR, Papadopoulou A, Thomas E, Tobias A, Price MJ, Meher S, Alfirevic Z, Weeks AD, Hofmeyr GJ, Gulmezoglu AM, Widmer M, Oladapo OT, Vogel JP, Althabe F, Coomarasamy A, Gallos ID. Uterotonic agents for first-line treatment of postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD012754. doi: 10.1002/14651858.CD012754.pub2. PMID 33232518
- [Derived] Abbas DF, Mirzazada S, Durocher J, Pamiri S, Byrne ME, Winikoff B. Testing a home-based model of care using misoprostol for prevention and treatment of postpartum hemorrhage: results from a randomized placebo-controlled trial conducted in Badakhshan province, Afghanistan. Reprod Health. 2020 Jun 5;17(1):88. doi: 10.1186/s12978-020-00933-8. PMID 32503556